CLINICAL TRIAL: NCT06940232
Title: Ubiquitin C-terminal Hydrolase L1 (UCH-L1) and Glial Fibrillary Acidic Protein (GFAP) as Acute Biomarkers for Prediction of Traumatic Brain Injury (TBI) in Children
Brief Title: Validating a Blood Test for the Detection of Traumatic Brain Injury in Children
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0423-24-EP
Record Dates: First submitted 2025-04-14; First posted 2025-04-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Traumatic Brain Injury
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Group 1 - Traumatic Brain Injury With Positive Head Computed Tomography Findings: Group 1 will be 110 participants who had a traumatic brain injury (TBI) with positive head computed tomography (HCT).
  Interventions: Diagnostic Test: Blood Test for Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) Acute Biomarkers
- Group 2 - Traumatic Brain Injury With Negative Head Computed Tomography Findings: Group 2 will be 110 participants with a known traumatic brain injury (TBI), but a negative head computed tomography (HCT).
  Interventions: Diagnostic Test: Blood Test for Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) Acute Biomarkers
- Group 3 - All Other Trauma Participants With No History of Head Injury: Group 3 will be 110 participants being treated for a traumatic injury with no history of head injury.
  Interventions: Diagnostic Test: Blood Test for Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) Acute Biomarkers

INTERVENTIONS:
Diagnostic Test: Blood Test for Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) Acute Biomarkers — All groups will have blood drawn per standard of care. Blood samples will be analyzed using Traumatic Brain Injury (TBI) cartridges for iSTAT Alinity device.

SUMMARY:
The primary objective of this study is to establish if Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) are predictive of computed tomography (CT) findings in pediatric traumatic brain injuries (TBI). The participant population is pediatric patients, ages 0 to less than 18 years old with a possible TBI or trauma-related injury who have blood drawn per standard of care in the emergency department. Blood samples will be analyzed using the i-STAT TBI cartridge (Abbott Laboratories, Abbott Park, IL, USA) by the Emergency Department charge nurse within one hour of collection of the blood sample. Clinical outcomes will be assessed via telephone interview with a parent at 3 and 6 months for all surviving TBI patients.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) estimates 3,000 deaths annually in children and youth from traumatic brain injury (TBI), 29,000 hospitalizations, and 400,000 emergency room visits . A prospective study lead by the Pediatric Emergency Care Applied Research Network (PECARN) reported that 35.5% of 40,000 children who presented with a mild TBI (Glasgow Coma Scale, GCS, 14-15) had a head computed tomography (CT) scan, of which only 0.9% were clinically significant, and 0.1% required neurosurgical intervention, which led to the development of an algorithm for the need for CT imaging in pediatric mild TBI. However, a large scale study of the National Hospital Ambulatory Care Medical Survey database from 2008-2015 did not show a decrease in children undergoing CT imaging. Thus, there is still a need for a more definitive means to predict intracranial injury to avoid radiation exposure in children.

In 2018, the US Food and Drug Administration (FDA) approved the first blood test to assess mild TBI for adults with suspected brain injury. A portable point-of-care platform was made available that could detect concentrations of serum and plasma concentrations of Glial Fibrillary Acidic Protein (GFAP) and Ubiquitin C-terminal Hydrolase L1 (UCH-L1) in 15 minutes to predict evidence of intra-cranial hemorrhage on CT. Although not yet FDA approved in children, some studies showed that GFAP and UCH-L1 were able to distinguish children with concussive symptoms from body trauma controls, while others showed significantly higher levels of GFAP, but not UCH-L1. These studies did not test the hypothesis of serum biomarkers for prediction of evidence of intracranial injury on cranial imaging. Thus, further studies are needed to determine if these biomarkers can be used in the pediatric population to predict degree of intracranial injury.

Investigators propose a prospective case-control study that is comprised of three groups: participants with mild TBI, Glasgow Coma Scale (GCS) 13-15, participants with moderate to severe TBI (GCS <13), and a control group that includes other trauma participants with no history of head injury. Patients under the age of 18 (0-17) who present to the emergency room in the setting of non-penetrating trauma will be screened. All patients with blood obtained for clinical purposes will be included in the study. Written consent for prospective follow-up will be obtained from parents prior to discharge from the hospital. Participant demographic and clinical information will be abstracted from chart review.

The aims of the study are to determine GFAP and UCH-L1 levels within 24 hours of head injury in children with moderate/severe TBI (GCS 3-12) compared to those with mild TBI (GCS 13-15) and trauma patients without clinical concern for TBI, to determine if serum GFAP and UCH-L1 levels are higher in children with TBI and an abnormal head CT scan compared to those with TBI and normal head CT scan, and to determine if higher serum GFAP and UCH-L1 are predictive of worse clinical outcomes 3 and 6 months after TBI via the Post-Concussion Symptom Inventory and the Pediatric Cerebral Performance Category Scale surveys.

ELIGIBILITY:
Inclusion Criteria:

* 0-17 years of age
* Presentation of non-penetrating trauma
* Blood draw within 24 hours of injury
* For TBI group: head CT or MRI obtained

Exclusion Criteria:

* Presentation to Children's Nebraska after 24 hours of injury
* 18 years of age or older

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under the age of 18 (0-17) who present to the emergency room in the setting of non-penetrating trauma and blood draw within 24 hours of injury will be screened. All participants who present as a trauma activation will automatically have blood drawn as part of the trauma protocol. Participants with head trauma who do not present as a trauma activation (i.e. arrived via private auto) will have labs drawn at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Serum Glial Fibrillary Acidic Protein Levels, an Acute Biomarker, Among Children With Traumatic Brain Injury and Control Groups | Within 24 hours of injury
  Serum Glial Fibrillary Acidic Protein (GFAP) levels measured with a i-STAT TBI cartridge within 24 hours of head injury will be compared in children with moderate/severe traumatic brain injury (TBI), Glasgow Coma Scale (GCS) 3-12, mild TBI (GCS 13-15) and trauma participants without clinical concern for TBI.
Comparison of Ubiquitin C-terminal Hydrolase L1 Levels, an Acute Biomarker, Among Children With Traumatic Brain Injury and Control Groups | Within 24 hours of injury
  Serum Ubiquitin C-terminal Hydrolase L1 (UCH-L1) levels measured with a i-STAT TBI cartridge within 24 hours of head injury will be compared in children with moderate/severe traumatic brain injury (TBI), Glasgow Coma Scale (GCS) 3-12, mild TBI (GCS 13-15) and trauma participants without clinical concern for TBI.
Comparison of Serum Glial Fibrillary Acidic Protein Levels, an Acute Biomarker, Between Children With Traumatic Brain Injury With Normal and Abnormal Head Computed Tomography Scan | Within 24 hours of injury
  Serum Glial Fibrillary Acidic Protein (GFAP) measured with a i-STAT TBI cartridge within 24 hours of traumatic brain injury (TBI) and a normal head computed tomography (CT) scan will be compared to levels in children with TBI and an abnormal head computed tomography (CT) scan.
Comparison of Ubiquitin C-terminal Hydrolase L1 Levels, an Acute Biomarker, in Children With Traumatic Brain Injury With Normal and Abnormal Head Computed Tomography Scan | Within 24 hours of injury
  Serum Ubiquitin C-terminal Hydrolase L1 (UCH-L1) levels in children with traumatic brain injury (TBI) and a normal head computed tomography (CT) scan will be compared to levels in children with (TBI) and an abnormal head computed tomography (CT) scan.
Comparison of Serum Glial Fibrillary Acidic Protein Levels, an Acute Biomarker, and Clinical Outcomes in Children With Traumatic Brain Injury Using Post-Concussion Symptom Inventory | 3 months and 6 months after traumatic brain injury
  Serum Glial Fibrillary Acidic Protein (GFAP) levels in children with traumatic brain injury (TBI) will be compared to clinical outcomes using the Post-Concussion Symptom Inventory. The Inventory rates 23 symptoms from 0 (none) to 6 (severe).
Comparison of Ubiquitin C-terminal Hydrolase L1 Levels, an Acute Biomarker, and Clinical Outcomes in Children With Traumatic Brain Injury Using Post-Concussion Symptom Inventory | 3 months and 6 months after traumatic brain injury
  Serum Ubiquitin C-terminal Hydrolase L1 (UCH-L1) levels in children with traumatic brain injury (TBI) will be compared to clinical outcomes using the Post-Concussion Symptom Inventory. The Inventory rates 23 symptoms from 0 (none) to 6 (severe).
Comparison of Serum Glial Fibrillary Acidic Protein Levels, an Acute Biomarker, and Clinical Outcomes in Children With Traumatic Brain Injury Using Pediatric Cerebral Performance Category Scale | 3 months and 6 months after traumatic brain injury
  Serum Glial Fibrillary Acidic Protein (GFAP) levels in children with traumatic brain injury (TBI) will be compared to clinical outcomes using the Pediatric Cerebral Performance Category Scale. This scale rates 5 functional categories from 1 (normal) to 6 (vegetative state).
Comparison of Ubiquitin C-terminal Hydrolase L1 Levels, an Acute Biomarker, and Clinical Outcomes in Children With Traumatic Brain Injury Using Pediatric Cerebral Performance Category Scale | 3 months and 6 months after traumatic brain injury
  Serum Ubiquitin C-terminal Hydrolase L1 (UCH-L1) levels in children with traumatic brain injury (TBI) will be compared to clinical outcomes using the Pediatric Cerebral Performance Category Scale. This scale rates 5 functional categories from 1 (normal) to 6 (vegetative state).

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lai, MD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Children's Nebraska, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No